CLINICAL TRIAL: NCT05422690
Title: A Phase II Single-center, Open-label, Single Arm Study of Induction Gemcitabine, Cisplatin and Durvalumab Followed by Gemcitabine, Cisplatin and Yttrium-90 (Y-90) Radioembolization for the Treatment of Locally Advanced Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: The Purpose of This Research Study is to See if Combining Gemcitabine, Cisplatin and Durvalumab Chemotherapy Treatments With a Direct Tumor Therapy Yittrium-90 (Y-90) Will Work Better Together to Shrink Tumors and Control Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U22-02-4670
Record Dates: First submitted 2022-05-27; First posted 2022-06-16 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Intervention Model Description: Treatments are repeated every 21 days. Chemotherapy will be administered on days 1 and 8 of the 21 day cycle. For the first two cycles, treatment will consist of three drugs, gemcitabine, cisplatin and Durvalumab.
  After these two cycles, the Durvalumab will be removed from the treatment plan and participants will continue on trial with gemcitabine and cisplatin alone for 6 additional cycles (8 total cycles, or 6 months total of treatment). During the 3rd and possibly the 4th cycle, these drugs will be given at a reduced dose as y-90 treatment to the tumors in your liver will also be given. The interventional team will administer y-90 during these cycles as either one dose during cycle 3, or two doses, one during cycle 3 and one during cycle 4 if there is too much cancer to treat all at once.
  The remaining cycles of treatment will be with gemcitabine and cisplatin by themselves.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- gemcitabine, cisplatin and Durvalumab chemotherapy with Yittrium-90 (Experimental): single arm - Induction Gemcitabine, Cisplatin and Durvalumab Triplet Chemotherapy followed by Gemcitabine, Cisplatin in combination with yttrium-90 (Y-90) Radioembolization
  Interventions: Drug: Induction Chemotherapy Triplet Therapy; Radiation: Concurrent Y-90 treatment; Drug: Consolidation Doublet Therapy:

INTERVENTIONS:
Drug: Induction Chemotherapy Triplet Therapy — Gemcitabine 1000 mg/m2, Cisplatin 25 mg/m2 infused on both day 1 and day 8 of a 21-day cycle. Durvalumab 1500 mg will be given on day 1 of each cycle.
Radiation: Concurrent Y-90 treatment — Patients will undergo a Y-90 treatment planning consultation by the treating interventional radiologist during cycle 1. One or two cycles (depending on tumor size) of cisplatin, 25 mg/m2 and gemcitabine 300 mg/m2 given on day 1 and day 8 in combination with Yttrium-90 (Y-90) microspheres which will be given on day 3-7 or day 10-21 at the discretion of the interventional radiologist, separated in time by at least 2 days from a chemo infusion during that cycle
Drug: Consolidation Doublet Therapy: — Gemcitabine 1000 mg/m2 and Cisplatin 25 mg/m2 given on days 1 and 8 of a 21-day cycle with durvalumab 1500 mg given on day 1 of each cycle for 3-5 additional cycles. For the cycle directly after Y-90, gemcitabine will be kept at a dose of 300 mg/m2 to minimize risk of toxicity.

SUMMARY:
The purpose of this research is to see if combining gemcitabine, cisplatin and Durvalumab chemotherapy treatments with a direct tumor therapy called Yittrium-90, will work better together to shrink the tumor and control cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females at least 18 years of age
* Histologically and/or cytologically confirmed iCCA that is previously untreated or, if systemic therapy has been rendered for prior disease, has been administered at least 6 months before the development of recurrent or de novo new sites of disease.
* Unresectable disease, as deemed by the Inova multidisciplinary tumor board (i.e. disease that cannot be safely resected with negative margins, leaving 2 adjacent segments of liver with intact portal venous and hepatic arterial inflow and intact biliary and hepatic venous outflow with the future liver remnant of sufficient volume to avoid postoperative liver insufficiency)
* Measurable disease per RECIST 1.1 at least 2 cm in size
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Noncirrhotic liver - patients should not have a preexisting diagnosis of cirrhosis either diagnosed via biopsy or with features consistent with cirrhosis on imaging (e.g. shrunken liver with nodularity consistent with cirrhosis). Child-Pugh score must be less than 5.
* No evidence of extrahepatic disease, except for regional adenopathy that would be resected as part of a standard oncologic surgical procedure
* Adequate organ function as indicated by the following laboratory values (Table 1)
* Ability to complete testing in the protocol
* Able and willing to consent to protocol

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* History of allogeneic organ transplantation.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled type 1 diabetes on an insulin regimen are eligible for the study.
  * Patients with vitiligo or alopecia.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients without an active autoimmune disease in the last 5 years may be included but only after consultation with the study physician.
  * Patients with diet controlled celiac disease.
* Current or recent use of immunosuppressive medication within 14 days before durvalumab initiation except if:

  * Intranasal, inhaled, topical or local steroid injections
  * Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or its equivalent.
  * Steroids as premedication for hypersensitivity reactions, (i.e. CT scan premedication).
* Child-Pugh B7 or greater cirrhosis
* Extrahepatic or perihilar cholangiocarcinoma
* Gallbladder cancer
* Pancreatic or ampullary cancer
* Portal vein thrombosis involving the main portal vein or first order right or left portal vein branches
* Extrahepatic disease, other than regional lymph nodes that would be removed at time of surgery as part of a routine oncologic procedure for iCCA
* Previous treatment with chemotherapy, intra-arterial or radiotherapy for iCCA is exclusionary, with the exception of adjuvant therapy with capecitabine which is allowed.
* Contraindication to durvalumab, gemcitabine, or cisplatin
* Active hepatitis B or C for which patients refuse treatment. Patients who are newly diagnosed with active disease as part of protocol screening and are agreeable to initiate on antiviral treatment are allowed to enroll.
* Contraindication found during work-up angiography, including significant lung shunting (lung dose >30 Gy for a single treatment or >50 Gy cumulative), or non-manageable extrahepatic deposition of technetium Tc 99m macroaggregated albumin on scintigraphy performed after planning angiography
* > 75% hepatic tumor burden
* Inability to protect non-target arteries to intestines or solid organs from radioembolization
* Serum albumin < 3 g/dL
* Serum bilirubin > 2 mg/dL, serum aspartate aminotransferase or alanine aminotransferase > 5 times upper limit of normal
* Concomitant illness that would prevent adequate patient assessment or in the investigators' opinion pose an added risk for study participants.
* Life-threatening intercurrent illness
* Anticipated poor compliance
* Prisoners or subjects who are involuntarily incarcerated
* Persons with decisional incapacity/cognitive impairment
* Any history or evidence of severe illness or any other condition that would make the patient, in the opinion of the investigator unsuitable for the study
* Subject is enrolled in a separate interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the objective response rate (ORR) at 6 months in patients with locally advanced, unresectable intrahepatic cholangiocarcinoma (iCCA) | 6 months
  Best response in terms of tumor shrinkage (by RECIST 1.1 criteria including complete + partial responses) obtained during protocol therapy.

SECONDARY OUTCOMES:
Assessing Progression Free Survival (PFS) | 48 months
  time from treatment initiation to disease progression, death or last patient contact
Hepatic Progression-Free Survival (HPFS) | 48 months
  time from treatment initiation to hepatic disease progression, death or last patient contact
Overall Survival (OS) | 48 months
  Time from treatment initiation to death due to any cause or last patient contact
Disease Control Rate (DCR) | 48 months
  Complete Response + Partial Response + Stable Disease (by RECIST 1.1 and mRECIST criteria) obtained during protocol therapy.
R0 resection rate | 6 months
  Rate of patients that achieve an R0 resection at 6 months.
treatment related impact on quality of life | 48 months
  Self-assessed metric of treatment-related impact on Quality of Life (QOL) as measured by the Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) questionnaire with measures of Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Hepatobiliary Cancer Subscale using a 5 point scale ((0) Not at all (1) A little bit; (2) Somewhat; (3) Quite a bit; (4) Very much). Better performance status, i.e. higher score, is associated with a higher quality of life.
safety and toxicity rate | 48 months
  Development of Treatment Toxicities (grade 3 non-hematologic toxicities persisting beyond 2 weeks despite best supportive care, any grade 3 hematologic toxicities, or any toxicity grade 4 or higher) assessed as per NCI's CTCAE v5.0 criteria.
rate of downstaging to surgery | 6 months
  Rate of downstaging to surgery that occurs during protocol therapy at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur A. Winer, MD, Principal Investigator — Inova Schar Cancer Institute
Locations (1):
- Keary Janet, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Saha SK, Zhu AX, Fuchs CS, Brooks GA. Forty-Year Trends in Cholangiocarcinoma Incidence in the U.S.: Intrahepatic Disease on the Rise. Oncologist. 2016 May;21(5):594-9. doi: 10.1634/theoncologist.2015-0446. Epub 2016 Mar 21. PMID 27000463
- [Background] Ribero D, Pinna AD, Guglielmi A, Ponti A, Nuzzo G, Giulini SM, Aldrighetti L, Calise F, Gerunda GE, Tomatis M, Amisano M, Berloco P, Torzilli G, Capussotti L; Italian Intrahepatic Cholangiocarcinoma Study Group. Surgical Approach for Long-term Survival of Patients With Intrahepatic Cholangiocarcinoma: A Multi-institutional Analysis of 434 Patients. Arch Surg. 2012 Dec;147(12):1107-13. doi: 10.1001/archsurg.2012.1962. PMID 22910846
- [Background] Si A, Li J, Xiang H, Zhang S, Bai S, Yang P, Zhang X, Xia Y, Wang K, Yan Z, Lau WY, Shi L, Shen F. Actual over 10-year survival after liver resection for patients with intrahepatic cholangiocarcinoma. Oncotarget. 2017 Jul 4;8(27):44521-44532. doi: 10.18632/oncotarget.17815. PMID 28562348
- [Background] Tarchi P, Tabrizian P, Prigoff J, Schwartz M. Outcomes of resection for solitary </=5 cm intrahepatic cholangiocarcinoma. Surgery. 2018 Apr;163(4):698-702. doi: 10.1016/j.surg.2017.09.058. Epub 2017 Dec 23. PMID 29277385
- [Background] Yeh CN, Hsieh FJ, Chiang KC, Chen JS, Yeh TS, Jan YY, Chen MF. Clinical effect of a positive surgical margin after hepatectomy on survival of patients with intrahepatic cholangiocarcinoma. Drug Des Devel Ther. 2014 Dec 17;9:163-74. doi: 10.2147/DDDT.S74940. eCollection 2015. PMID 25552905
- [Background] Lang H, Sotiropoulos GC, Fruhauf NR, Domland M, Paul A, Kind EM, Malago M, Broelsch CE. Extended hepatectomy for intrahepatic cholangiocellular carcinoma (ICC): when is it worthwhile? Single center experience with 27 resections in 50 patients over a 5-year period. Ann Surg. 2005 Jan;241(1):134-43. doi: 10.1097/01.sla.0000149426.08580.a1. PMID 15622001
- [Background] Mazzaferro V, Gorgen A, Roayaie S, Droz Dit Busset M, Sapisochin G. Liver resection and transplantation for intrahepatic cholangiocarcinoma. J Hepatol. 2020 Feb;72(2):364-377. doi: 10.1016/j.jhep.2019.11.020. PMID 31954498
- [Background] De Martin E, Rayar M, Golse N, Dupeux M, Gelli M, Gnemmi V, Allard MA, Cherqui D, Sa Cunha A, Adam R, Coilly A, Antonini TM, Guettier C, Samuel D, Boudjema K, Boleslawski E, Vibert E. Analysis of Liver Resection Versus Liver Transplantation on Outcome of Small Intrahepatic Cholangiocarcinoma and Combined Hepatocellular-Cholangiocarcinoma in the Setting of Cirrhosis. Liver Transpl. 2020 Jun;26(6):785-798. doi: 10.1002/lt.25737. PMID 32090444
- [Result] Ilyas SI, Khan SA, Hallemeier CL, Kelley RK, Gores GJ. Cholangiocarcinoma - evolving concepts and therapeutic strategies. Nat Rev Clin Oncol. 2018 Feb;15(2):95-111. doi: 10.1038/nrclinonc.2017.157. Epub 2017 Oct 10. PMID 28994423
- [Result] Akateh C, Ejaz AM, Pawlik TM, Cloyd JM. Neoadjuvant treatment strategies for intrahepatic cholangiocarcinoma. World J Hepatol. 2020 Oct 27;12(10):693-708. doi: 10.4254/wjh.v12.i10.693. PMID 33200010
- [Result] Labib PL, Davidson BR, Sharma RA, Pereira SP. Locoregional therapies in cholangiocarcinoma. Hepat Oncol. 2017 Oct;4(4):99-109. doi: 10.2217/hep-2017-0014. Epub 2017 Nov 17. PMID 29367874
- [Result] Hyder O, Marsh JW, Salem R, Petre EN, Kalva S, Liapi E, Cosgrove D, Neal D, Kamel I, Zhu AX, Sofocleous CT, Geschwind JF, Pawlik TM. Intra-arterial therapy for advanced intrahepatic cholangiocarcinoma: a multi-institutional analysis. Ann Surg Oncol. 2013 Nov;20(12):3779-86. doi: 10.1245/s10434-013-3127-y. Epub 2013 Jul 12. PMID 23846786
- [Result] Kuhlmann JB, Euringer W, Spangenberg HC, Breidert M, Blum HE, Harder J, Fischer R. Treatment of unresectable cholangiocarcinoma: conventional transarterial chemoembolization compared with drug eluting bead-transarterial chemoembolization and systemic chemotherapy. Eur J Gastroenterol Hepatol. 2012 Apr;24(4):437-43. doi: 10.1097/MEG.0b013e3283502241. PMID 22261548
- [Result] Sommer CM, Kauczor HU, Pereira PL. Locoregional Therapies of Cholangiocarcinoma. Visc Med. 2016 Dec;32(6):414-420. doi: 10.1159/000453010. Epub 2016 Dec 5. PMID 28229076
- [Result] Han K, Ko HK, Kim KW, Won HJ, Shin YM, Kim PN. Radiofrequency ablation in the treatment of unresectable intrahepatic cholangiocarcinoma: systematic review and meta-analysis. J Vasc Interv Radiol. 2015 Jul;26(7):943-8. doi: 10.1016/j.jvir.2015.02.024. Epub 2015 Apr 18. PMID 25899049
- [Result] Pillai K, Akhter J, Chua TC, Shehata M, Alzahrani N, Al-Alem I, Morris DL. Heat sink effect on tumor ablation characteristics as observed in monopolar radiofrequency, bipolar radiofrequency, and microwave, using ex vivo calf liver model. Medicine (Baltimore). 2015 Mar;94(9):e580. doi: 10.1097/MD.0000000000000580. PMID 25738477
- [Result] Yang L, Shan J, Shan L, Saxena A, Bester L, Morris DL. Trans-arterial embolisation therapies for unresectable intrahepatic cholangiocarcinoma: a systematic review. J Gastrointest Oncol. 2015 Oct;6(5):570-88. doi: 10.3978/j.issn.2078-6891.2015.055. PMID 26487951
- [Result] Zhen Y, Liu B, Chang Z, Ren H, Liu Z, Zheng J. A pooled analysis of transarterial radioembolization with yttrium-90 microspheres for the treatment of unresectable intrahepatic cholangiocarcinoma. Onco Targets Ther. 2019 Jun 7;12:4489-4498. doi: 10.2147/OTT.S202875. eCollection 2019. PMID 31239717
- [Result] White J, Carolan-Rees G, Dale M, Patrick HE, See TC, Bell JK, Manas DM, Crellin A, Slevin NJ, Sharma RA. Yttrium-90 Transarterial Radioembolization for Chemotherapy-Refractory Intrahepatic Cholangiocarcinoma: A Prospective, Observational Study. J Vasc Interv Radiol. 2019 Aug;30(8):1185-1192. doi: 10.1016/j.jvir.2019.03.018. Epub 2019 Jun 27. PMID 31255499
- [Result] Weigt J, Malfertheiner P. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. Expert Rev Gastroenterol Hepatol. 2010 Aug;4(4):395-7. doi: 10.1586/egh.10.45. PMID 20678012
- [Result] Shroff RT, Javle MM, Xiao L, Kaseb AO, Varadhachary GR, Wolff RA, Raghav KPS, Iwasaki M, Masci P, Ramanathan RK, Ahn DH, Bekaii-Saab TS, Borad MJ. Gemcitabine, Cisplatin, and nab-Paclitaxel for the Treatment of Advanced Biliary Tract Cancers: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):824-830. doi: 10.1001/jamaoncol.2019.0270. PMID 30998813
- [Result] Edeline J, Touchefeu Y, Guiu B, Farge O, Tougeron D, Baumgaertner I, Ayav A, Campillo-Gimenez B, Beuzit L, Pracht M, Lievre A, Le Sourd S, Boudjema K, Rolland Y, Boucher E, Garin E. Radioembolization Plus Chemotherapy for First-line Treatment of Locally Advanced Intrahepatic Cholangiocarcinoma: A Phase 2 Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):51-59. doi: 10.1001/jamaoncol.2019.3702. PMID 31670746
- [Result] Cheng B, Villalobos A, Sethi I, Wagstaff W, Galt J, Brandon D, Schuster DM, Bercu Z, Majdalany B, Kokabi N. Determination of Tumor Dose Response Thresholds in Patients with Chemorefractory Intrahepatic Cholangiocarcinoma Treated with Resin and Glass-based Y90 Radioembolization. Cardiovasc Intervent Radiol. 2021 Aug;44(8):1194-1203. doi: 10.1007/s00270-021-02834-0. Epub 2021 Apr 22. PMID 33890170
- [Result] Camacho JC, Kokabi N, Xing M, Prajapati HJ, El-Rayes B, Kim HS. Modified response evaluation criteria in solid tumors and European Association for The Study of the Liver criteria using delayed-phase imaging at an early time point predict survival in patients with unresectable intrahepatic cholangiocarcinoma following yttrium-90 radioembolization. J Vasc Interv Radiol. 2014 Feb;25(2):256-65. doi: 10.1016/j.jvir.2013.10.056. PMID 24461131